CLINICAL TRIAL: NCT03223766
Title: Phase IV Clinical Trial of Proton Therapy in Pediatric Cancer
Brief Title: Evaluation of Proton Therapy in Pediatric Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SJPROTON1
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Tumor
Keywords: Proton therapy; Long-term effects
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Participants will be those enrolled to receive proton therapy on other protocols at SJCRH on or after November 18, 2015.

SUMMARY:
This is a Phase IV clinical trial observing and evaluating the safety of proton therapy in children. Protocol therapy is not being done as part of this clinical trial. The radiation targeting, planning, prescribed dose, fractionation, schedule, and use of other forms of therapy will be done per other therapeutic protocols at St. Jude Children's Research Hospital (SJCRH) at the discretion of the treating physicians associated with those trials.

DETAILED DESCRIPTION:
For the clinical trial being described in this registration, participants will be observed to collect data for baseline assessment of disease and patient characteristics. This will be done before proton therapy on other trials followed by serial standard-of-care clinical assessments to evaluate acute and late complications, disease control, treatment-related mortality, and overall survival.

PRIMARY OBJECTIVE:

* To estimate the incidence of radiation associated grade 3 and grade 4 non-hematologic toxicities at 1, 3, 5, and 10 years in a radiated region specific manner after the initiation of proton therapy.

SECONDARY OBJECTIVES:

* To estimate the incidence of necrosis, vasculopathy, and symptomatic and permanent neurologic deficits at 1, 3, 5, and 10 years after the initiation of proton therapy in children treated for central nervous system (CNS) tumors in an irradiated region directed manner.
* To estimate the incidence of treatment-related mortality at 5 and 10 years after the initiation of proton therapy.
* To estimate the incidence of subsequent malignancies at 5 and 10 years after the initiation of proton therapy in an irradiated region directed manner.
* To estimate the incidence of fracture and osteonecrosis at 1, 3, 5, and 10 years after the initiation of proton therapy in children treated for musculoskeletal tumors in an irradiated region directed manner.

ELIGIBILITY:
Inclusion Criteria:

* The patient is planned for treatment or has been treated with proton therapy at St. Jude Children's Research Hospital on or after November 18, 2015.

Exclusion Criteria:

* Patients who are currently pregnant will not be enrolled in the study as radiation has teratogenic or abortifacient effects. In the rare case that a patient was previously pregnant as a young adult, the patient will be considered eligible for enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants will be patients at St. Jude Children's Research Hospital. They must meet eligibility criteria to be considered for enrollment. No one group (based on gender, race or ethnicity) will be targeted or excluded.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2037-07 (Estimated); Study Completion 2037-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of radiation-associated non-hematologic toxicities | From baseline through 10 years
  All Grade 3 and Grade 4 non-hematologic toxicities will be reviewed to determine attribution to proton therapy given in other clinical trials at SJCRH and the number reported.

CONTACTS AND LOCATIONS:
Overall Officials: John T. Lucas, Jr., MS, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols